CLINICAL TRIAL: NCT01088568
Title: Randomized, Prospective Comparison of the Outcome of TICL and Q Value Customized LASIK for the Correction of Myopia With Astigmatism
Brief Title: Randomized, Prospective Comparison of the Outcome of Toric Implantable Contact Lens (TICL) and Q-LASIK for the Correction of Myopia With Astigmatism
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Wenzhou Medical University (Other)
Collaborators: Staar Surgical Company (Industry)
Responsible Party: Qinmei Wang MD, Eye hospital of Wenzhou Medical College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20091231
Record Dates: First submitted 2010-03-16; First posted 2010-03-17 (Estimated); Last update posted 2010-03-17 (Estimated); Status verified 2009-10

CONDITIONS: Myopia; Astigmatism
Keywords: Keratomileusis, laser in situ; Phakic Intraocular Lenses; myopia; astigmatism; Implantable Collamer Lens, Toric
MeSH Terms: conditions — Myopia; Astigmatism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TICL group (Experimental)
  Interventions: Procedure: the implantation of toric implantable collamer lens
- LASIK group (Active Comparator)
  Interventions: Procedure: customized laser-assisted in situ keratomileusis

INTERVENTIONS:
Procedure: the implantation of toric implantable collamer lens — perform the implantation of toric implantable collamer lens for both eyes
  Other Names: TICL
  Arms: TICL group
Procedure: customized laser-assisted in situ keratomileusis — perform Q-factor customized laser-assisted in situ keratomileusis for both eyes
  Other Names: Q-factor customized LASIK
  Arms: LASIK group

SUMMARY:
The objective is to conduct a contralateral prospective clinical study to compare the safety, efficacy, and quality of vision of the STAAR Surgical Co. Toric Implantable Contact Lens TICL) versus Custom Laser Vision Correction (Q-LASIK) in human eyes for the correction of myopia with astigmatism.

ELIGIBILITY:
Inclusion Criteria:

* Age: 21-45 years old
* Documented stable refraction for at least 1 year
* (-3.0 to -8.0D of myopia with -1.0 to -4.0D of astigmatism or SE from -3.5 to -10D
* BSCVA: 20/20 or better
* Pupil diameter: smaller than 7mm under mesopic condition
* Contact lens discontinued 3 weeks and 1 week for hard and soft wearers respectively

Exclusion Criteria:

* Evidence of progressive or acute disease
* Evidence of connective tissue disease or clinically significant atopic disease
* ACD less than 2.8mm from endothelium
* ECC less than 2200 cells/mm2
* Narrow angle of anterior chamber
* Residual stromal thickness less than 280 microns

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2007-11; Primary Completion 2008-12 (Actual); Study Completion 2010-03 (Estimated)

PRIMARY OUTCOMES:
Comparing the efficacy, predictability, stability and safety of TICL versus Q-LASIK | 1week, 1,3,6 months

SECONDARY OUTCOMES:
Comparing wavefront aberrometry of TICL vs Q-LASIK Comparing contrast sensitivity of TICL vs Q-LASIK Comparing patient satisfaction of TICL vs Q-LASIK | 1, 3, 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Qin Mei Wang, Study Director — Eye hospital of Wenzhou Medical College
Locations (1):
- Eye hospital of Wenzhou Medical College, Wenzhou, Zhejiang, China

REFERENCES:
- [Background] Sanders DR. Matched population comparison of the Visian Implantable Collamer Lens and standard LASIK for myopia of -3.00 to -7.88 diopters. J Refract Surg. 2007 Jun;23(6):537-53. doi: 10.3928/1081-597X-20070601-02. PMID 17598571
- [Background] Sanders D, Vukich JA. Comparison of implantable collamer lens (ICL) and laser-assisted in situ keratomileusis (LASIK) for low myopia. Cornea. 2006 Dec;25(10):1139-46. doi: 10.1097/ICO.0b013e31802cbf3c. PMID 17172886
- [Background] Sanders DR, Vukich JA. Comparison of implantable contact lens and laser assisted in situ keratomileusis for moderate to high myopia. Cornea. 2003 May;22(4):324-31. doi: 10.1097/00003226-200305000-00009. PMID 12792475